CLINICAL TRIAL: NCT07356141
Title: Apple Watch Assessment of Dental Stress in Special Needs Treatment
Brief Title: Monitoring Occupational Dental Stress Using Apple Watch
Status: Not yet recruiting | Type: Observational
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Shlomo Elbahary, Clinical Associate Professor, University of Illinois at Chicago
Other Study IDs: STUDY2025-1178
Record Dates: First submitted 2026-01-12; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Increased Heart Rate
MeSH Terms: conditions — Tachycardia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patient with special needs
- Patients with capability

SUMMARY:
* This study will enroll 10 dental students (primary subjects) and up to 200 patients (secondary subjects), approximately 10 special-needs and 10 non-special-needs encounters per student, totaling about 200 treatment sessions.
* Students will wear an Apple Watch to continuously monitor heart rate (HR) during routine care. The Apple Watch contains built-in physiological sensors that automatically record heart rate and heart rate variability. These data are stored locally in the Apple Health app on a study-designated iPhone that is assigned for the research and handled solely by the Principal Investigator (PI). No real-time transmission or cloud-based sharing occurs during data recording. No additional apps, accounts, or third-party software are used. At designated intervals, the PI will use the health app's built-in "Export Health Data" function on the study iPhone. This function generates a ZIP file containing an export.xml file with sensor-recorded data. The PI will then upload the ZIP file from the study iPhone directly to a secure, university-approved UI Box Health Data Folder designated for the study. No research account will be set up for this purpose.
* A trained observer will record start/stop timepoints of procedure phases (e.g., seating, anesthesia start, operative phase, dismissal) to align with HR signals and will document only minimal patient variables needed for analysis: behavior/cooperation score (e.g., Frankl), sedation status, and broad procedure category (e.g., preventive, restorative, surgical).
* Each dental student will complete the Perceived Stress Questionnaire (PSQ) only once at the beginning of the study to stablish a baseline measure of stress. The Questionnaire takes approximately 5 minutes to complete. Students do not need to complete the PSQ for each patient encounter. Student HR data and permitted minimal patient variables will be coded and de-identified, stored securely in UI Box Health Data Folder, and analyzed to compare special-needs vs non-special-needs encounters and to evaluate associations between student HR and the listed patient factors. No additional patient identifiers or PHI will be collected beyond what is specified above.

ELIGIBILITY:
Inclusion Criteria:

* Students (primary subjects) inclusion criteria: After IRB approval, non-supervisory staff or research team members will invite potential participants via UIC email/listservs. Interested students will be screened confirming: (a) good academic standing and current clinical assignment, (b) routine provision of care to both special-needs and non-special needs patients during the data-collection window, (c) willingness to wear an Apple Watch during sessions and complete baseline/end PSQ, and (d) absence of medical/dermatologic conditions that would preclude safe/accurate wrist-worn monitoring. Screening and consent occur privately and outside evaluative contexts.
* Patient (secondary subjects) Inclusion criteria: Patients will be screened at the point of care when already scheduled with a participating student. A pre-visit check confirms capacity to consent (or availability of a legally authorized representative/parent/guardian). For minors and/or special needs patients, LAR permission will be obtained in addition to assent to the research. The following criteria will be considered:
* Minors and/or Special-needs patients who are scheduled for standard clinical care with a participating student during the study period may be enrolled as secondary subjects provided that their parent/guardian or legally authorized representative (LAR) grants permission during the consent process and the patient assents to the research when appropriate.
* Adult Patients with capacity who are scheduled for standard clinical care with a participating student during the study period may be enrolled as secondary subjects provided that are willing to provide informed consent.
* Willing to allow an observer and collection of minimal visit-level variables (behavior/cooperation score, sedation status, broad procedure category).
* Patients and/or their parent(s), guardian(s), or legally authorized representative(s) providing consent must be able to understand and communicate in English.

Exclusion Criteria:

* Students (primary subjects) Exclusion criteria:
* Not assigned to patient-care rotations during the study window.
* Known dermatologic, cardiovascular, neurologic, or other medical conditions that would interfere with safe or accurate HR monitoring or tolerability of a wrist device.
* Unwilling or unable to provide consent or follow procedures.
* Patients (secondary subjects) Exclusion criteria:
* Declines consent/permission/assent or withdraws at any time.
* Prisoners or individuals under custodial supervision.
* Pregnant women

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Primary Subjects - Dental Students:
  Ten (10) dental students enrolled at the University of Illinois Chicago (UIC) College of Dentistry will participate. These students will provide routine clinical care to both special needs and non-special needs patients as part of their standard educational and clinical responsibilities.
  Secondary Subjects - Patients Receiving Care:
  Approximately 200 patients will be observed during these clinical sessions, including both special needs patients treated in the Inclusive Care Clinic (ICC) and non-special needs patients treated in other UIC dental clinics. Special needs patients and/or their legally authorized representatives (LARs) will provide consent, and, when appropriate, patients will provide assent.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Heart rate changes in dental students during dental procedures | During each dental treatment session per session

CONTACTS AND LOCATIONS:
Locations (1):
- University of Illinois Chicago (UIC) College of Dentistry, Chicago, Illinois, United States